CLINICAL TRIAL: NCT02229188
Title: Games to Overcome Late Life Depression
Acronym: GOLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Pat Arean, Professor, Psychiatry and Behavioral Sciences, University of Washington
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY00001751
Record Dates: First submitted 2014-08-26; First posted 2014-09-01 (Estimated); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Major Depressive Disorder
Keywords: Depression; mood; cognitive training
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Biological Evolution

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Problem Solving Therapy (Active Comparator): Problem Solving Therapy is an evidence-based behavioral treatment for late life depression proven effective with different geriatric groups including ambulatory; medically ill; older adults with executive dysfunctions; and more recently, low-income, disabled older adults.
  Interventions: Behavioral: Problem Solving Therapy
- Evolution (Experimental): Evolution is a plasticity intervention in the form of a video driving game that targets the cognitive conflict network.
  Interventions: Behavioral: Evolution
- Words (Placebo Comparator): Words is a challenging crosswords type of game that will serve as the placebo comparator to Evo.
  Interventions: Behavioral: Words

INTERVENTIONS:
Behavioral: Problem Solving Therapy — Problem solving therapy is an evidence based behavioral intervention for late life depression. It consist of 8 weekly session of talk therapy, whereby the therapist helps the patient solve problems that are thought to be causing depressive symptoms.
  Other Names: PST
  Arms: Problem Solving Therapy
Behavioral: Evolution — Evo is a video game that has therapeutic elements targeting the cognitive control network. Impairment in this neural network is associated with a specific subtype of late life depression that puts people at risk for poor response to SSRIs. Evo is built from a research grade training paradigm that has shown to induce improvements in this network in healthy older adults
  Other Names: Neuroracer; Evo; Project: Evolution
  Arms: Evolution
Behavioral: Words — Words is a cognitively challenging crossword/word search type of video game that will serve as the control condition for the second phase of this project
  Arms: Words

SUMMARY:
This is a pilot study divided into two phases. IN phase 1 (completed) participants will be randomized to receive 8 weeks of Problem Solving Therapy (PST) alone or 8 weeks of a cognitive training game called, Evolution (Evo) plus clinical management. In Phase 2 (now recruiting), participants will be randomized to Evo, PST, and a different cognitive training program called Words. Words is similar to Evo in that it is an adaptive training program and includes case management. IN both studies participants will be assessed for clinical and functional magnetic resonance imaging (fMRI) outcomes at baseline, 4 weeks and 8 weeks.

DETAILED DESCRIPTION:
Evo is a computer game that targets parts of the brain (i.e. the cognitive control network) that we think may be associated with depressive symptoms. This study is exploratory and will inform future hypotheses the research team will test in subsequent research.

ELIGIBILITY:
Inclusion Criteria:

1. Between 60-80 years of age
2. Meets criteria for Major Depressive Disorder
3. Hamilton Depression Rating Scale (HDRS) of 20 or greater
4. Mini Mental State Exam score of 24 or greater
5. Can speak and read English
6. Able to physically participate in the research protocol (e.g.: is not suffering from a terminal or highly disabling illness)
7. Can participate in MRI scans
8. Able to provide written informed consent

Exclusion Criteria:

1. History of psychosis, mania, or currently using or abusing illicit drugs or alcohol
2. Diagnosis of dementia
3. Taking cognitive enhancers
4. Change in or newly began taking psychiatric medication within the last 6 months
5. Pacemaker
6. Metal in the body that cannot be removed
7. Color blind
8. Movement disorder that prevents participation -

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Change in depression over time | weeks 0, 4, 8, 24
  Hamilton Depression Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Arean, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Department of Psychiatry and Behavioral Sciences, Seattle, Washington, United States

REFERENCES:
- [Derived] Anguera JA, Gunning FM, Arean PA. Improving late life depression and cognitive control through the use of therapeutic video game technology: A proof-of-concept randomized trial. Depress Anxiety. 2017 Jun;34(6):508-517. doi: 10.1002/da.22588. Epub 2017 Jan 3. PMID 28052513